CLINICAL TRIAL: NCT06540846
Title: Deep Learning for Histopathological Classification and Prognostication of Gynaecologic Smooth Muscle Tumours
Acronym: STUMP
Status: Recruiting | Type: Observational
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Other Study IDs: IB2023-STUMP
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Stump
Keywords: algorithm; diagnostic; pronostic
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — digitalized slides
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- STUMP cohort: Smooth muscle tumors of the uterus that do not fit the diagnostic criteria of benignity (such as leiomyomas) or malignancy (such as leiomyosarcomas) : smooth muscle tumor of uncertain malignant potential
  Interventions: Other: No intervention
- Leiomyoma-leiomyosarcoma: Smooth muscle tumors of the uterus that do fit the diagnostic criteria of benignity (such as leiomyomas) or malignancy (such as leiomyosarcomas)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention since this is an observational study

SUMMARY:
Smooth muscle tumors of the uterus that do not fit the diagnostic criteria of benignity (such as leiomyomas) or malignancy (such as leiomyosarcomas) are called STUMP (smooth muscle tumor of uncertain malignant potential). A potential solution to this problem could be the application of predictive models using artificial intelligence (AI) to aid in the histopathological classification and prognosis of gynecological smooth muscle tumors. Deep learning using convolutional neural networks represents a specific class of machine learning, in which predictive models are trained by considering small groups of pixels in digital images and iteratively identifying salient features. In this study, we aim to develop deep learning models capable of accurately subclassifying and predicting the prognosis of gynecological smooth muscle tumors, based on histopathological features of hematoxylin and eosin (H&E) slides. The aim is to develop a diagnostic and prognostic algorithm to help pathologists better classify and diagnose uterine smooth muscle tumors and predict their clinical course.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of uterine smooth muscle tumors (leiomyomas, smooth muscle tumors of uncertain malignancy and leiomyosarcomas), registered in the RRePS database and/or treated at Institut Bergonié or one of the participating centers.
* Histopathological material available (kerosene blocks and/or slides).
* The follow-up (outcome) is required for each LMS/ STUMP.

Exclusion Criteria:

* na

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — only uterin tumors
Study Population: - Uterine smooth muscle tumors: leiomyomas, smooth muscle tumors of uncertain malignancy and leiomyossarcomas.
Sampling Method: Non-Probability Sample
Enrollment: 392 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Develop deep learning models that can accurately subclassify gynaecologic smooth muscle tumours | throughout the conduct of the study - an expected average of 6 months after data collection
  This project aims to improve the diagnosis and prognosis of gynecologic smooth muscle tumors, including leiomyomas (LM), leiomyosarcomas (LMS), and smooth muscle tumors of uncertain malignant potential (STUMP). In detail, a workflow comprising 2 stages will be developed to automatically classify GSMT subtypes from whole-slide images and to predict progression-free survival for patients in the LMS and STUMP groups, thereby providing clinicians with a more effective tool to improve workflow quality.

SECONDARY OUTCOMES:
Develop a prognostic tool for STUMP | 6 months after receiving the data.
  Develop a model to predict progression-free survival for STUMP group based on the features extracted from Whole Slide Images.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Bergonie, Bordeaux, France